CLINICAL TRIAL: NCT02690155
Title: Real-world Comparative Effectiveness of Rivaroxaban Versus VKA
Acronym: RIVA-F
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18734
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation (NVAF); Prevention; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban: NVAF patients who were initiated on rivaroxaban for stroke prevention
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- VKA (Vitamin K antagonist): NVAF patients who were initiated on VKA for stroke prevention
  Interventions: Drug: VKA (Vitamin K antagonist)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — As prescribed by treating physicians
  Groups: Rivaroxaban
Drug: VKA (Vitamin K antagonist) — As prescribed by treating physicians
  Groups: VKA (Vitamin K antagonist)

SUMMARY:
To obtain a better understanding on the comparative effectiveness of rivaroxaban versus VKA(Vitamin K antagonist) for stroke prevention in patients with NVAF(non-valvular atrial fibrillation) in a real-life setting

ELIGIBILITY:
Inclusion Criteria:

* NVAF(non-valvular atrial fibrillation) will be defined as the occurrence of 2 or more inpatient or outpatient claims with ICD(International Classification of Disease)-9 427.31 as the diagnosis code at any time in the patient's data history prior to inclusion
* Patients will be required to have 180 days of enrollment for the assessment of baseline characteristics
* CHA2DS2-Vasc score ≥2 during the 180 days prior to index rivaroxaban use baseline period (CHA2DS2-Vasc: Diabetes mellitus; S2: prior Stroke or TIA or Thromboembolism; V: Vascular disease; A: Age 65-74 years; Sc: Sex category)

Exclusion Criteria:

* Patients <18 years of age
* Patients with valvular AF (Atrial fibrillation)
* Pregnancy
* Malignant cancers
* Transient cause of AF
* Patients with venous thromboembolism (pulmonary embolism or deep vein thrombosis)
* Patients with major surgery defined as hip or knee replacement
* Prescriptions of oral anticoagulants (OACs) (apixaban, warfarin, dabigatran, rivaroxaban) before index date
* Prescription of more than one OAC on the index date
* Patient with any of the events defined in the composite endpoint

  * Fatal bleeding
  * Fatal Stroke/Myocardial infarction
  * Intracranial hemorrhage
  * Ischemic stroke
  * Myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation (NVAF)
Sampling Method: Non-Probability Sample
Enrollment: 38831 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Hospitalization Events (composite endpoint) | Within 2 years of starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- New York, New York, United States